CLINICAL TRIAL: NCT06652529
Title: First in Human Phase 1 Dose Escalation and Expansion Clinical Trial to Evaluate the Safety, Pharmacokinetics and Antitumor Activity of Intravenous AROG4-01 in Patients With Advanced Solid Tumors
Brief Title: Phase 1 Dose Escalation and Expansion to Evaluate AROG4-01 in Patients With Advanced Solid Tumors
Acronym: AROG4-01-01
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aromics Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AROG4-01-01
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumors (Phase 1); Mesothelioma; Colorectal Carcinoma; Ovarian Cancer; NSCLC (Advanced Non-small Cell Lung Cancer)
Keywords: Phase I; AROG4-01; mesothelioma; solid tumors; NSCLC; ovarian cancer; colorectal cancer; dose escalation
MeSH Terms: conditions — Mesothelioma; Colorectal Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: This clinical trial is divided into two parts: dose escalation (part A), and dose expansion (part B). In part A (dose escalation), patients will be treated with AROG4-01 at different doses, starting at 9 mg/m2. Escalation to next dose levels will occur following the Safety Review Committee meeting for the most recently completed cohort.
  The MTD decided as per part A (dose escalation) will be used for part B (dose expansion).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): Four dose levels will be tested. If there are no safety concerns, dose escalation may continue with up to two additional dose levels
  Interventions: Drug: AROG4-01

INTERVENTIONS:
Drug: AROG4-01 — AROG4-01 will be administered as IV infusions in biweekly dosing interval. The first dosing day will be Day 1, 28 days cycle.
  Other Names: Dose level 2; Dose level 3; Dose level 4; Dose level 5; Dose level 6; dose level 1
Drug: AROG4-01 — AROG4-01 will be administered as IV infusions in biweekly dosing interval. The first dosing day will be Day 1, 28 days cycle.
  This study is an open label, Phase 1 dose escalation trial with two expansion cohorts. The study consists of two parts:
  * Part A: Dose escalation in patients with advanced solid tumors. Approximately 8 to 20 patients in total will be enrolled in part A, covering up to 6 dose levels.
  * Part B: At the dose expansion phase, AROG4-01 two cohorts of ten patients with advanced solid tumor each will be recruited. One cohort of patients with advanced MPM (cohort 1) and a second cohort of patients with other solid tumors (cohort 2).

SUMMARY:
The goal of this clinical trial is to learn if drug AROG4-01 is safe in patients with solid tumors who have no available treatment alternative. Different doses will be tested in order to identify the most suitable one. Once it is identiffied, up to 20 patients will be treated with that dose, to check if thye get clinical benefit.

Participants will: receive intravenous administrations of ARG4-01 twice weekly, and visit the clinic twice every week for checkups and tests.

DETAILED DESCRIPTION:
This study is an open label, Phase 1 dose escalation trial with two expansion cohorts to investigate the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary antitumor activity of AROG4-01 in patients with mesothelioma and other advanced solid tumors.

This clinical trial is divided into two parts: dose escalation (part A), and dose expansion (part B).

Dose escalation In the present trial, patients will be enrolled sequentially into escalating dose cohorts, and will continue receiving AROG4-01 until disease progression, unacceptable toxicity, withdrawal of consent or otherwise as specified in the investigational medicinal product (IMP) discontinuation criteria.

Patients in a dose cohort will receive AROG4-01 as intravenous (IV) administrations at the same dose in a dosing interval of twice a week, four weeks (equal to one cycle) consecutively without interruption, except when necessary to manage adverse events (AEs).

Six cohorts at escalating dose levels are envisaged. Dose escalation may continue beyond, until the recommended for part B dose, which will be the recommended for phase 2 dose (RP2D), can be defined based on safety, preliminary efficacy, PK and PD data, based on the recommendations of the Safety Review Committee (SRC). The RP2D is defined as the recommended for phase 2 dose, but two cohorts will be treated as part of the phase 1 expansion with that particular dose, in order to get more safety and efficacy data.

Escalation to the next dose level will occur following the SRC meeting for the most recently completed cohort. In considering the appropriate dose level for the next cohort the following will be applied:

* The maximum dose increment will be limited to 100% if patients of a given cohort experience one Grade ≥ 2 AE during the DLT period or if at least one patient decreases >10% weight.
* The maximum dose increment will be limited to 50% if a patient of a given cohort experiences one DLT during the DLT period.

If the prior circumstances do not occur, dose escalation will continue at higher increments (not exceeding three times prior dose level), as determined by the SRC.

Extension phase At the dose expansion part, two cohorts of patients with advanced solid tumor each will be recruited. One cohort of patients with advanced MPM (cohort 1) and a second cohort of patients with other solid tumors (cohort 2). Patients will be treated with AROG4-01 at the RP2D of AROG4-01 resulting from part A.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 18 years or older, with a diagnosis (histology or citology) of advanced (unresectable or metastatic) solid tumor for which there is no curative therapy, has progressed on SOC treatment or for whom SOC is no longer an option. In part B patients will be included in different cohorts according to the histology (mesothelioma vs. non-mesothelioma).
2. Evaluable (part A) or measurable disease (part B) as per RECIST v1.1 (part A) or mRECIST v1.1. (part B). Progressive disease to the on or following the last line of antitumor treatment.
3. ECOG performance status ≤ 2.
4. Life expectancy ≥12 weeks.
5. Hematology and clinical chemistry laboratory parameters within acceptable ranges.
6. Adequate organ function as defined below:

   * Hemoglobin ≥9 g/dL
   * Neutrophil count ≥1.000x10/mcL
   * Platelets ≥100.000/mcL
   * Total bilirubin ≤1,5 x Upper Limit of Normal (ULN) (unless Gilbert's Disease)
   * AST (SGOT)/ALT (SGPT) ≤ 2,5 x institutional ULN (or ≤ 5X ULN in the presence of liver metastases)
   * Creatinine ≤1.5 mg/dL and creatinine CL ≥40 mL/min (calculated using the Cockcroft-Gault formula)
7. Adequate coagulation profile as defined below:

   * INR≤ 1,5
   * aPTT ≤ 1,5 x ULN
   * Serum or urine negative pregnancy test for women with childbearing potential.
8. No previous antitumor treatment (radiation therapy, systemic treatment, or surgery) in the previous 28 days and current adverse events from them ≤ grade 1.

Exclusion Criteria:

1. Systemic anti-cancer therapy within 4 weeks prior to study admission.
2. Radiation therapy within 4 weeks prior to study entry.
3. Any major surgery within 4 weeks before first dose of study treatment No major surgery must be planned during the trial expected treatment. receiving study treatment. Participants with recent surgery with only local anesthesia may be included.
4. Non-malignant systemic disease including cerebrovascular accident, myocardial infarction in the last 6 months, unstable angina pectoris, unstable cardiac arrhythmia, New York Heart Association (NYHA) Class III or IV heart failure, coagulation abnormalities and clinically significant pulmonary compromise, .
5. Left ventricular ejection fraction below institutional normal limits.
6. Patients with symptomatic central nervous system (CNS) primary tumor or metastases (including leptomeningeal carcinomatosis). Patients with documented treated CNS metastases stable for at least 4 weeks may be enrolled at the discretion of the investigator.
7. Breast feeding, pregnancy or not willing to adopt safe contraceptive measures by the patient or the patient's partner, to become pregnant during treatment or within 6 months after the end of treatment.
8. Patients with active uncontrolled infection or known to be serologically positive for human immunodeficiency virus (HIV), hepatitis B (except HbsAc after vaccination) or hepatitis C infection.
9. Any other diseases or medical condition that may interfere with the planned treatment, compliance, or place the patient at risk if participating in the study, at investigator criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of AROG4-01 | 12 months
  To evaluate the safety and tolerability of AROG4-01 in adult patients with advanced solid tumors, including determination of the main DLT associated to AROG4-01.
  To assess the MTD (RP2D) defined as the highest dose at which no more than one in six patients experience a AROG4-01-related DLT. DLTs will be evaluated after the first treatment cycle.

SECONDARY OUTCOMES:
To assess the preliminary antitumor activity of AROG4-01 monotherapy as measured by Overall Response Rate (ORR) according to standard criteria (RECIST 1.1 [18] or mRECIST v1.1 | 24 months
  • To assess progression-free survival (PFS) in patients with mesothelioma and other advanced solid tumors.
To characterize the PK of AROG4-01. | 24 months
  Cmax
To characterize the PK of AROG4-01 | 12 months
  half-life

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aubets E, J Felix A, Garavis M, Reyes L, Avino A, Eritja R, Ciudad CJ, Noe V. Detection of a G-Quadruplex as a Regulatory Element in Thymidylate synthase for Gene Silencing Using Polypurine Reverse Hoogsteen Hairpins. Int J Mol Sci. 2020 Jul 16;21(14):5028. doi: 10.3390/ijms21145028. PMID 32708710
- [Background] 19- Phan, A. T., & Patel, D. J. (2005). "RNA tetraplexes, structures and functions." Biochemistry, 44(2), 639-649. doi:10.1021/bi048804m
- [Background] Simon, J. S., et al. (2018). "Hairpin structures near G-quadruplexes can modulate G4 stability and drug binding." Nature Communications, 9, 4621. doi:10.1038/s41467-018-07055-8
- [Background] Rhodes D, Lipps HJ. G-quadruplexes and their regulatory roles in biology. Nucleic Acids Res. 2015 Oct 15;43(18):8627-37. doi: 10.1093/nar/gkv862. Epub 2015 Sep 8. PMID 26350216
- See also: Company website — https://www.aromics.es/en/
- Available data/document: Study Protocol — https://www.aromics.es/en/